CLINICAL TRIAL: NCT02833220
Title: The Effects of Single-Pulse Transcranial Magnetic Stimulation on the Autonomic Nervous System in Healthy Adults
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: TMS and BP
Record Dates: First submitted 2016-07-11; First posted 2016-07-14 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: blood pressure; heart rate variability; single-pulse transcranial magnetic stimulation; non-invasive brain stimulation
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy volunteers: * Healthy adults between the ages of 18-65 are eligible.
  * Participants will receive non-invasive brain stimulation by way of single-pulse transcranial magnetic stimulation to the motor cortex
  Interventions: Device: Single-Pulse Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Single-Pulse Transcranial Magnetic Stimulation — Single-pulse Transcranial Magnetic Stimulation activates neurons within the cortex of the brain by way of electromagnetic induction. This causes a small, focused electric field to become present in the brain, which activates the neurons.

SUMMARY:
The purpose of this study is to determine the effects of TMS on the ANS. The investigator will determine whether single-pulse TMS of the primary motor cortex in the dominant hemisphere in healthy, young adults will affect 1) heart rate and heart rate variability, 2) blood pressure and 3) baroreflex function. This study is foundational in that it will begin to characterize how single-pulse TMS affects the ANS in healthy adults.

DETAILED DESCRIPTION:
The overall purpose of this study is to investigate the effects of TMS on the ANS. Specifically; the investigator aim to determine if single-pulse TMS of the primary motor cortex in the dominant hemisphere in healthy, young adults will significantly affect 1) heart rate and heart rate variability, 2) blood pressure and 3) baroreflex function.

The first purpose of this study is to measure alterations in sympathetic and parasympathetic activation in response to TMS. To do this, we will measure HRV immediately after single-pulse TMS. The second purpose is to investigate the changes in blood pressure in response to TMS and to determine whether the baroreflex, a critical modulator of blood pressure, is inhibited by TMS.

Aim 1: To determine if single-pulse TMS of the primary motor cortex will significantly alter heart rate variability. We hypothesize that single-pulse TMS of the primary motor cortex will elicit an acute decrease in heart rate and result in improved heart rate variability indicated by a significantly decreased LF power and increased HF power.

Aim 2: To determine if single-pulse TMS of the primary motor cortex will significantly alter blood pressure and baroreflex sensitivity (BRS). We hypothesize that single-pulse TMS of the primary motor cortex will elicit an acute decrease in blood pressure by inhibiting the baroreflex.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers between 18-65 years old

Exclusion Criteria:

* pregnant or breastfeeding women
* previous episodes of seizures or fainting
* any implanted metal in their head
* history of migraines
* history of psychiatric disorder (e.g. depression, anxiety, ADHD, bi-polar disorder)
* currently taking medications that may alter autonomic function (e.g. blood pressure medication, depression medication)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-01; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in Blood Pressure during the intervention as compared to baseline | Change from baseline
  It is possible that blood pressure is changing when the single-pulse transcranial magnetic stimulation is being delivered.

SECONDARY OUTCOMES:
Change in Heart Rate Variability from baseline | Change from baseline
  Heart rate variability is a non-invasive measurement of the activity of the parasympathetic nervous system

CONTACTS AND LOCATIONS:
Overall Officials: Manda L Keller-Ross, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No